CLINICAL TRIAL: NCT00284778
Title: A Randomized Cost-minimization Trial Comparing Pemetrexed (Alimta®) Versus Docetaxel (Taxotere®) as Second Line Treatment in Advanced Non Small Cell Lung Cancer (NSCLC): Study 05-06 of Groupe Français de Pneumo-Cancérologie (GFPC).
Brief Title: Pharmaco-economic Study of a Second Line Treatment in Advanced Non Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Collaborators: Groupe Francais De Pneumo-Cancerologie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I05026
Record Dates: First submitted 2006-01-31; First posted 2006-02-01 (Estimated); Last update posted 2025-07-24 (Actual); Status verified 2010-03

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: lung cancer; second line treatment; cost-minimization trial; Pharmaco-economic study; docetaxel; pemetrexed
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Pemetrexed; Docetaxel

ARMS (2):
- ALIMTA (Experimental)
  Interventions: Drug: Alimta®
- Docetaxe (Active Comparator)
  Interventions: Drug: Taxotere®

INTERVENTIONS:
Drug: Alimta®
  Arms: ALIMTA
Drug: Taxotere®
  Arms: Docetaxe

SUMMARY:
The indication of chemotherapy of 2nd line treatment in advanced non small cell lung cancer is now well established. The two treatments of reference are pemetrexed (alimta) and docetaxel (taxotere). Effectiveness and toxicity of the two drugs are largely documented in the literature.

Economic analyses are currently one of the criteria used in medical decision, beside effectiveness, quality of life and toxicities.

However, Economical comparison shows significant variations in the acquisition costs of the two drugs. Consequently, it appears interesting to carry out a randomized prospective study with on exclusive economical criteria of judgment.

As there is no difference in the effectiveness between the two treatments, a cost-minimization analysis will be carried out to appreciate the ratio benefit/risks from an economical point of view (payer).

DETAILED DESCRIPTION:
The main objective of this trial is of to compare, economically, the use of pemetrexed (alimta®) in 2nd line chemotherapy in advanced non-small cell lung cancer versus docetaxel (taxotere®).

150 patients will be selected for this trial which, after checking the eligibility criteria, will be randomized in two arms:

* Arm A: Taxotere 75 mg/m² every 3 weeks.
* Arm B : Alimta 500 mg/m² every 3 weeks.

Inclusion assessment.

* Clinical signs
* Blood cell count, renal and hepatic function (within 8 days)
* Chest X ray, CT scan or MRI scan, abdominal echography, and/or abdominal scan (within 28 days)
* Brain scan, bone scintigraphy and/or bone x ray (within 28 days)
* Bronchial endoscopy (within 28 days)
* EKG, echocardiography according to history

Follow-up assessment.

1. At each cycle

   * Clinical signs
   * Blood cell count at D1, D8, D15
   * Creatinine, serum electrolytes (K+, Ca++ ), SGOT, SGPT, total bilirubin, LDH, alkaline phosphate, total protein and albumin, EKG, Chest X-ray at D1
2. Follow-up each 2 months till PD
3. End of trial: Complete tumor assessment
4. Each objective response may be confirm 4 weeks later

Length ot the study.

* Patients in each arm will be treated until progression or toxicity or decision to stop the trial.
* Responder patient will be treated until 6 cycles. The follow-up assessment will be carried out each 2 months.

Response assessment. According to RECIST criteria.

Resource consumption.

1. Recording of volumes:

   * All the medication quantities will be recorded in mg. The chemotherapeutic products will be recorded in mg. All the concomitant treatments : RHO, anti-emetics, growth factors, antibiotics or adverse event treatments will be notified.
   * Hospitalizations for treatment and their categories ( inpatient, outpatient, home based treatment) will be noted.
   * All the hospitalizations for adverse events will be recorded (and their category). Grade 1-2 adverse events will be notified in the case report form. Hospitalizations for disease complications or progressions, curative or palliative radiation will be recorded.
2. Cost calculation :

   * All hospitalisations will be valued by DRGs or day hospitalisation prices, according to the country. Ambulatory care will be valued by appropriate country prices. The drug price will be done by pharmaceutical companies.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proved stage IV or pleural stage III NSCLC (neoplastic pleurisy confirmed).
* Metastatic relapses allowed if asymptomatic.
* Progressive disease during or after a standard first line platinum-based chemotherapy (without taxotere or alimta)
* Only one chemotherapeutic line including adjuvant and neo adjuvant treatment.
* Irradiation allowed if < 25% bone medulla . It may be ended 2 weeks before the second line treatment.
* At least one measurable target lesion according to recist criteria in non previously irradiated area.
* Performance status <=2
* Age between 18 and 70 years
* Life expectancy > 12 weeks.
* Normal hepatic function
* Normal renal function
* Normal serum calcium
* Absolute neutrophil count>1.5 gigal/l,platelets>100 gigal/l,haemoglobin>9.0 g/dl
* Written informed consent

Exclusion Criteria:

* SCLC, bronchioli-alveolar and neuro-endocrine carcinoma.
* Symptomatic brain metastases.
* Superior vena cava syndrome.
* Uncontrolled fluid retention in the third space (pleural or ascitic collection)
* Prior chemotherapy without platin
* Other concomitant diseases: heart failure, angina pectoris, tachyarrythmia, recent myocardial infarction, active infections.
* Peripheral neuropathy grade ≥ 2.
* Past or concomitance of another cancer except baso-cellular carcinoma of the skin or in situ cervical carcinoma.
* Hypersensitivity to docetaxel or polysorbate 80.
* Unability or unwillingness to take folic acid, vitamin B12 supplementation or corticosteroids.
* Pregnancy or breast feeding.
* Follow-up of the patient impossible.
* Prisoners

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2006-02; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alain Vergnenegre, MD, Principal Investigator — CHU Limoges; Christos Chouaid, MD, Study Chair — Hôpital Saint Antoine; Paris
Locations (18):
- France (18):
  - Service de Pneumologie, CHU Angers, Angers
  - Service de pneumologie; Centre Hospitalier d'Annecy, Annecy
  - Service de Pneumologie; Centre Hospitalier, Beauvais
  - Service de Pneumologie ; Centre hospitalier, Charleville-Mézières
  - Service de Pneumologie; Centre Hospitalier, Draguignan
  - Service de Pathologie Respiratoire; CHU de Limoges, Limoges
  - Service de Pneumologie; Hôpital de la Croix Rousse, Lyon
  - Service de Pneumologie-Neurologie ; Centre Hospitalier F. Quesnay, Mantes-la-Jolie
  - Département des Maladies Respiratoires ; Hôpital Sainte Marguerite, Marseille
  - Service de Pneumologie et Réanimation ; Hôpital Hôtel Dieu - Paris, Paris
  - Service de Pneumologie - Hôpital St Antoine, Paris, Paris
  - Service de Pneumologie ; Hôpital saint Antoine, Paris, Paris
  - Service de Pneumologie-Allergologie; Centre Hospitalier Général, Périgueux
  - Service de Pneumologie; CHG de Roanne, Roanne
  - Clinique Pneumologique; Hôpital Charles Nicolle, Rouen
  - Service de Pneumologie; Hôpital Bois Guillaume, Rouen
  - Service d'Oncologie Médicale; Clinique Sainte Marguerite, Toulon
  - Service de Pathologie Respiratoire; Hôpital d'Instruction des Armées Sainte-Anne, Toulon Naval

REFERENCES:
- [Result] Vergnenegre A, Corre R, Berard H, Paillotin D, Dujon C, Robinet G, Crequit J, Bota S, Thomas P, Chouaid C; 0506 GFPC Team. Cost-effectiveness of second-line chemotherapy for non-small cell lung cancer: an economic, randomized, prospective, multicenter phase III trial comparing docetaxel and pemetrexed: the GFPC 05-06 study. J Thorac Oncol. 2011 Jan;6(1):161-8. doi: 10.1097/JTO.0b013e318200f4c1. PMID 21150465